CLINICAL TRIAL: NCT03694340
Title: Optimization of Cochlear Implant MAP-parameters in Children, Reprogramming Based on Active Co-operation
Brief Title: Optimization of Cochlear Implant MAP-parameters in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VGRFOU-247791
Record Dates: First submitted 2018-09-28; First posted 2018-10-03 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Cochlear Implants; Evoked Potentials, Auditory; Child; Disabilities Hearing; Deafness; Hearing
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Intervention Model Description: Single-case research design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Re-programming of cochlear implant (Other): The cochlear implant is programmed with a new MAP based on behavioral measurements of T- and C-levels and used by the participant for 4 months before follow up.
  Interventions: Other: Re-programming of cochlear implant

INTERVENTIONS:
Other: Re-programming of cochlear implant — New MAP based on behavioral T- and C-levels

SUMMARY:
This project will complete a long-term follow up for children that have received cochlear implants (CI) early in life and had their CI's programmed based on objective measurements.

At Sahlgrenska University Hospital in Gothenburg, generally, all younger children (0-3 years), the last ten years, had their CI's programmed based on objective measurements. The programming of the CI carried out during the first year after the surgical insertion is done on the foundation of the objective measurements and is generally what the child will live with thereafter. This method also seem to be close to other clinics in Sweden and the rest of the world, however, there are no specific guidelines regarding the how the programming of the CI is to be carried out on small children. To this date there are no studies, to our knowledge, that have confirmed the validity of using these objective measurements and if it is the best for the child. We therefore aim to do a long term follow up on children that have received CI and programmed this way, and study if there would be beneficial to redo the programming when the child is old enough to actively participate.

The aim with this project is evaluate how suitable it is to mainly use objective measurements when programming the cochlear implant and, in addition to this, examine if the children's hearing can be improved if the programming is based on the behavioral measurements of sound when the children are old enough to participate in such. It will examine what happens with the end result if the programming foundation differentiates from one another; if there are any measurable differences in hearing skills.

The result from this project expects to generate knowledge that is highly important for those working with small children receiving CI's, and by extension it will benefit the children that rely on this device in there every day life.

DETAILED DESCRIPTION:
Cochlear implants (CI) enable hearing for persons who otherwise would have been deaf. A CI substitutes the sensory cells in the cochlea and stimulates the auditory nerve directly with weak electrical pulses. For children born deaf, or become deaf at an early age, prompt detection of this condition is important to since it enables the possibility of an early implantation of the CI and facilitates the child's development of a spoken language. When it comes to detecting deafness in newborns, Sweden has a well-functioning and widespread hearing screening program for infants, permitting children born deaf, or with severe hearing impairments, to be discovered very early. In general, children that are born deaf can get a CI implanted at about one year of age, if there are no other contraindications. Internationally it has become increasingly common for implants to be inserted at even lower ages, sometimes even as young as five months of age.

For small children who receive CI's at an early age it is not possible to perform measurements based on the child making subjective assessments of how the sound is perceived when the electrical stimulation is altered through the implant. Also, small children cannot judge and report back the quality of the sound. Instead, objective measurements are commonly used since they do not require the active participation of the child, along with observations of the child and how it spontaneously reacts to the sound stimulation. A common objective measurement is to find the lowest level of electrical stimulation required to obtain a response from the auditory nerve, i.e. the electrically evoked action potential (ECAP) threshold. The CI manufacturer Cochlear Ltd has developed an automatic system for this measurement. Based on such measurements, as the automatic ECAP-measurement, the electrical stimulation from the implant can adjusted to the so-called MAP, where the minimum and maximum stimulation levels (T- respectively C-levels) are set for each individual electrode on the implant to create the dynamic range of electrical stimulation. This MAP then becomes the basis for the child's ability to perceive sound.

Clinically, today (at Sahlgrenska University Hospital, Gothenburg, Sweden) a basic programming of the MAP is performed based on ECAP measurements, after which adjustment of only the overall level is carried out based on the child's reactions. However, no subjective measurement is made regarding threshold levels of stimulation through the implant or that the child actually perceives medium sound equally across the different channels. When the child can participate in sound field audiometry, adjustments of the MAP settings are made to get a straight audiogram, but basically, the children continue to use the setting based on the ECAP measurement. Adult patients with acquired deafness receiving CI are managed in a different manner than the children. The programming of the implant for adults is based on subjective measurements of how stimulation via individual electrodes is perceived. By measuring thresholds for individual electrodes, i.e. minimum audible stimulation (T-levels) and levels where stimulation is immediately below unpleasant strong (C-levels), then the MAP is programmed with an individual dynamic range for each electrode.

To our knowledge no previous study have explored how the MAP based on an ECAP measurement endures over time or if a re-programming should be carried out when the child reliably can participate in behavioral measurements, which is about seven years of age in terms of measuring T-levels. Studies have shown that there is a correlation between ECAP-thresholds and T- and C-levels for people who can participate actively. However, the relationship is relatively weak and some researchers have even considered it too weak for ECAP thresholds to be the basis for programming the implant. However, in most clinics, these thresholds are used as a basis for programming CI to small children.

Several of those who work with programming the MAP in small children claims to witness an adaptation in sensitivity of the auditory nerve to the applied stimulation; indicating that the results of the objective measurement could gradually change if there is an alternation in stimulation levels. However, there are no studies at this time that neither confirm nor deny this.

The aim of this project is to investigate and clarify how children who receive CI at an early age should be monitored and to evaluate the objective ECAP measurement as a basis for setting stimulation levels. It also aims to investigate if there is any change in the result of the ECAP measurement after adjustment has been made in the MAP. After completion of the study, the goal is to offer a better and more knowledge-based (re-) habilitation for children who receive CI's, for whom there are currently no definite guidelines for programming and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Cochlear implant by Cochlear Ltd type: CI24RE or newer
* Received cochlear implant before three years of age
* Have carried out hearing tests with tones and speech recognition

Exclusion Criteria:

* Malformation of the cochlea

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in speech perception | Performed at baseline and 4 months after intervention
  Sound field hearing test performed with a pre-recorded speech material consisting of everyday sentences.
Change in tone threshold | Performed at baseline and 4 months after intervention
  Sound field hearing test performed with tones to determine hearing thresholds.
Behavioral T-thresholds | Performed at intervention
  Behavioral measurements of the T-levels that constitutes the the lower level of the dynamic range when programming the cochlear implant (setting the MAP).
Behavioral C-thresholds | Performed at intervention
  Behavioral measurements of the C-levels that constitutes the upper level of the dynamic range when programming the cochlear implant (setting the MAP).
Change in automatically recorded electrical evoked action potential thresholds | Performed at baseline and 4 months after intervention
  The measurement used for programming the cochlear implant if not behavioral measurements are feasible (e.g. small children).

SECONDARY OUTCOMES:
Change in results from "Children's Home Inventory for Listening Difficulties" questionnaire | Performed at baseline and 4 months after intervention
  The questionnaire "Children's Home Inventory for Listening Difficulties" assesses the subjective effect on the child's hearing of the re-programming of the cochlear implant. The questionnaire refers both the participant (the child) and the caregiver separately, and consists of 15 questions of different everyday hearing situation. Each question is answered on a rating scale of 1 - 8; a higher grading indicates better hearing (i.e. better outcome). The result is presented as a mean of all the ratings for the participant and the caregiver, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Magnusson, PhD, Principal Investigator — Sahlgrenska University Hospital, Region Västra Götaland
Locations (1):
- Göteborgs Universitet, Institute of Neuroscience and Physiology, Section of Rehabilitation and Clinical Neuroscienses, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roland JT Jr, Cosetti M, Wang KH, Immerman S, Waltzman SB. Cochlear implantation in the very young child: Long-term safety and efficacy. Laryngoscope. 2009 Nov;119(11):2205-10. doi: 10.1002/lary.20489. PMID 19507225
- [Background] de Vos JJ, Biesheuvel JD, Briaire JJ, Boot PS, van Gendt MJ, Dekkers OM, Fiocco M, Frijns JHM. Use of Electrically Evoked Compound Action Potentials for Cochlear Implant Fitting: A Systematic Review. Ear Hear. 2018 May/Jun;39(3):401-411. doi: 10.1097/AUD.0000000000000495. PMID 28945656
- [Background] Abbas PJ, Brown CJ, Shallop JK, Firszt JB, Hughes ML, Hong SH, Staller SJ. Summary of results using the nucleus CI24M implant to record the electrically evoked compound action potential. Ear Hear. 1999 Feb;20(1):45-59. doi: 10.1097/00003446-199902000-00005. PMID 10037065
- [Background] Botros A, van Dijk B, Killian M. AutoNR: an automated system that measures ECAP thresholds with the Nucleus Freedom cochlear implant via machine intelligence. Artif Intell Med. 2007 May;40(1):15-28. doi: 10.1016/j.artmed.2006.06.003. Epub 2006 Aug 22. PMID 16920343
- [Background] Plant K, Law MA, Whitford L, Knight M, Tari S, Leigh J, Pedley K, Nel E. Evaluation of streamlined programming procedures for the Nucleus cochlear implant with the Contour electrode array. Ear Hear. 2005 Dec;26(6):651-68. doi: 10.1097/01.aud.0000188201.86799.01. PMID 16378000